CLINICAL TRIAL: NCT00829946
Title: Effects of Resistance Strength Training on Functional Capacity and Well Being of Anorexic Patients; A Randomized Controlled Trial
Brief Title: Effects of Resistance Strength Training on Functional Capacity and Well Being of Anorexic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Alejandro Lucia, Universidad Europea de Madrid, Madrid, Spain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R-0034/08
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Anorexia
Keywords: Strength training; Anorexia; Girls; Quality of life; Functional mobility
MeSH Terms: conditions — Anorexia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Experimental)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — Participants in the intervention group were enrolled in two training sessions per week for 12 weeks. The core portion of the training session consisted of 11 strength exercises engaging the major muscle groups, i.e. bench press, shoulder press, leg extension, leg press, leg curl, abdominal crunch, low back extension, arm curl, elbow extension, seated row and lateral pull-down. For each exercise, the participants performed one set of 8-15 repetitions (total of ~ 20s duration) with resting periods of 1-2 min between exercises. The load was gradually increased as the strength of each child improved, i.e. from 20-30% of 6 repetition maximum (6RM) at the start of the program to 50-60% of 6RM at the end. Participants also performed isometric contractions of large muscle groups (6 sets of 3 repetitions each, 20-30s duration per repetition) with their own body weight (for lower body exercises) or barbells (1-3kg) for upper body.

SUMMARY:
The purpose of the present randomized controlled trial was to determine the effects of a 3-month resistance training program (2 sessions/week) on the functional mobility and muscle function, muscular dynamic strength, body composition and quality of life of young anorexic outpatients (≤16 years). The investigators also assessed cardiorespiratory variables of clinical significance such as peak oxygen uptake.

DETAILED DESCRIPTION:
A total of 22 outpatients [20 female (Tanner stage II-IV), 2 male (Tanner stage IV); age range: 12-16 years] were finally eligible and thus participated in the study.

Participants in the intervention group were enrolled in two training sessions per week for 12 weeks. Each session lasted 60-70 min and started at ~11:30 a.m., after the intra-hospital psychotherapy session. The program was individually supervised, i.e. one instructor for every three patients.

Each session started and ended with a low intensity 10-15min warm-up and cool-down period respectively, consisting of stretching exercises involving all major muscle groups. The core portion of the training session consisted of 11 strength exercises engaging the major muscle groups, i.e. bench press, shoulder press, leg extension, leg press, leg curl, abdominal crunch, low back extension, arm curl, elbow extension, seated row and lateral pull-down. For each exercise, the participants performed one set of 8-15 repetitions (total of ~ 20s duration) with resting periods of 1-2 min between exercises. The load was gradually increased as the strength of each child improved, i.e. from 20-30% of 6 repetition maximum (6RM) at the start of the program to 50-60% of 6RM at the end. Stretching exercises of the muscles involved in the previous exercises were performed during the rest periods (21).

Participants also performed isometric contractions of large muscle groups (6 sets of 3 repetitions each, 20-30s duration per repetition) with their own body weight (for lower body exercises) or barbells (1-3kg) for upper body.

Outcome measures:

* Anthopometry
* Cardiorespiratory fitness
* Muscular strength
* Functional mobility
* Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of restrictive anorexia nervosa
* Age ≤ 16 years
* Undergoing intra-hospital psychotherapy and dietary counseling (two visits per week) in this Hospital
* Body mass index > 14.0 kg/m2

Exclusion Criteria:

* None

Max Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Quality of life
Anthropometry
Functional mobility

SECONDARY OUTCOMES:
Muscular strength
Cardiorespiratory fitness